CLINICAL TRIAL: NCT02821468
Title: Evaluation of the Evolution of Imaging Markers of Cartilage Degradation in Patients With Knee Osteoarthritis Receiving DROGLICAN: a Pilot Study
Brief Title: Evaluation of the Evolution of Imaging Markers of Cartilage Degradation in Patients With Knee Osteoarthritis Receiving DROGLICAN
Acronym: DRIP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bioiberica (Industry)
Collaborators: Artialis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CL/BIO/2015-005 V5
Record Dates: First submitted 2016-06-06; First posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Droglican (Experimental): Chondroitin Sulfate 1,200mg + Glucosamine Hydrochoride 1,500mg
  Interventions: Drug: Droglican; Drug: Paracetamol or oral NSAIDs excluding COX2 inhibitors
- Control (Experimental): Untreated arm
  Interventions: Drug: Paracetamol or oral NSAIDs excluding COX2 inhibitors

INTERVENTIONS:
Drug: Droglican — Combined Chondroitin Sulfate 1200 mg + Glucosamine Hydrochloride 1500 mg
  Arms: Droglican
Drug: Paracetamol or oral NSAIDs excluding COX2 inhibitors

SUMMARY:
A previous multicenter trial led by Bioiberica S.A. has confirmed the efficacy and safety of DROGLICAN for the treatment of osteoarthritis (OA) in patients with severe pain. The MOVES study was a phase IV, double blind, randomized and non-inferiority trial to compare the efficacy and safety of a fixed dose combination of glucosamine hydrochloride (GH) + chondroitin sulfate (CS) (DROGLICAN) versus celecoxib in patient with symptomatic knee OA with moderate to severe pain. This study concluded that both drugs reduced the WOMAC Pain subscale by 50% without significant difference between groups. Further, there was no difference in all secondary outcomes assessing patient's pain, functional capacity, stiffness, inflammation, joint swelling, effusion, and overall quality of life.

This new exploratory trial is aimed to evaluate the beneficial effect of DROGLICAN on the good health of the cartilage of patients suffering of knee osteoarthritis as revealed by qualitative assessment of cartilage biochemical composition in vivo.

DETAILED DESCRIPTION:
This study is a post-marketing, open, exploratory, multicenter trial with 2 parallel-groups of patients suffering from knee OA. Investigators will be private or public hospital rheumatologists, general practitioners, or articular disease specialists located in Belgium.

After evaluation by the investigator during a control visit or via on site-patient registry, potential participants will be asked to perform an inclusion visit (V1). During this visit, the investigator will assess the eligibility of the patients. Eligible patients will sign an informed consent. The investigator will make a general evaluation (demography, medical history, OA history, OA medication history, concomitant medications including "rescue treatments") and a pain evaluation. Synovial fluid will be collected in case of knee swelling.

Blood samples will be collected in a preselected clinical laboratory for future biomarkers analyses.

Patients will be asked to perform an MRI exam within 20 days following the inclusion visit and representing the MRI at baseline. A standard X-ray will be performed at the same imaging site if the last X-ray available is not responding to high quality standard.

For DROGLICAN arm, patients will be given investigational medicinal product (IMP) for a 6-month period via the hospital pharmacy where image acquisition will be performed. IMP intake will begin right after baseline MRI acquisition. Study arm attribution will be determined according to the order of enrolment at each investigating site and using a randomization list.

All study subjects (receiving DROGLICAN or untreated control) will be allowed to take paracetamol and oral NSAIDs excluding COX2 inhibitors to relief knee pain. Patients will be asked to use these "rescue medications" only when needed during the trial, beginning by Paracetamol (up to 3g/day) and NSAIDs as a second-line medication, and will be told to reduce their use if they do not feel the need for them. The use of rescue treatments during the month prior to each visit will be recorded by the investigator in a Case Report Form (CRF). All other treatments for osteoarthritis will be forbidden during the course of the study.

Patients will return for consultation after 6 month (V2) and 12 months (V3). At each visit, the investigator will make a general evaluation, and will record concomitant medications including rescue medications, adverse events and drop-outs.

For DROGLICAN arm, compliance to the IMP will be assessed by counting unused capsules within the investigation kit brought back by the patient. At V2, patients will be given IMP for the next 6 months. Patients will be asked to return to the investigator all unused capsules of IMP at the next visit.

Blood samples and synovial fluid (if applicable) will be collected for future biomarkers analyses. MRI will be done at 6 months (V2) and optionally at 12 months (V3). Finally, an optional X-ray might be performed at V3 depending on the result of the interim analysis.

Monthly phone calls will be made by the investigator to assess and encourage patient's compliance (for DROGLICAN arm), to record potential adverse event, new concomitant treatment and/or drop-off.

Patients' clinical data will be recorded at each visit in a CRF.

ELIGIBILITY:
Inclusion Criteria:

* Femorotibial knee OA (Uni- or bilateral)
* Responding to clinical and radiological criteria of American College of Rheumatology (ACR)
* Symptomatic for more than 6 months in the most painful knee
* Radiological K&L grade II-III in radiographs from less than 12 months
* Moderate-to-severe knee pain: knee pain score evaluated on Visual Analogue Scale (VAS) (0-100) ≥ 40 over the last 24 hours at the inclusion visit (the most painful knee is considered)
* Able to follow the instructions of the study
* Having signed an informed consent

Exclusion Criteria:

Related to the OA pathology

* Recent trauma (< 1 month) of the knee responsible of the symptomatic knee
* Concurrent articular disease interfering with the evaluation of OA and/or pain such as articular dysplasia, aseptic osteonecrosis, acromegaly, Paget's disease, hemophilia, hemochromatosis, chondromatosis, villonodular synovitis of the knee, seronegative spondyloarthropathy, rheumatoid arthritis, gouty arthritis , infectious arthritis, radiculalgia in the lower limbs, arteritis, etc.
* Radiological K&L grade I or IV
* Prosthesis in the target knee

Related to treatments

* Analgesics to manage OA knee pain 24h before inclusion visit
* Corticosteroids injection in the target knee in the month preceding inclusion
* Hyaluronan injection in the target knee in the last 6 months
* Oral corticotherapy ≥ 5mg/day in the last 3 months
* Symptomatic slow-acting drugs (SYSADs) treatment (Chondroitin, diacerein, glucosamine, soy and avocado unsaponifiables) in the last 3 months
* An anticipated need for any OA related medication for the duration of the trial (Corticosteroids or hyaluronan injection, Oral corticotherapy, Arthroscopy, analgesics other than the authorized rescue treatments) which are forbidden during the trial
* Arthroscopy in the last 6 months
* Patients with known allergy to CS, GH, or intolerance to rescue treatment (Paracetamol and NSAIDs)
* Patients with allergy to shellfish

Related to associated diseases

* Severe and uncontrolled diseases (liver or renal failure, lung/heart severe disease, tumor, HIV….)
* Anticipated need for any surgical or other invasive procedure during the trial including prosthesis in the target knee Related to patients
* Artialis (study coordinator) or Bioiberica (Sponsor) 's employees
* Participation to a therapeutic clinical trial in the last 3 months
* Under guardianship or judicial protection
* Pregnancy, breastfeeding, planned conception
* Women without menopause or tubal ligation and without contraception

Related to MRI

* Unable to receive gadopentetate contrast agent injection because of contraindications:
* Acute or chronic severe renal insufficiency (a glomerular filtration rate < 30 mL/min/1.73m2); or
* Acute renal insufficiency of any severity due to the hepato-renal syndrome or in the peri-operative liver transplantation period.
* Known anaphylactic reactions to Gadolinium or related substances
* Risk groups for MRI scanning due to magnetic field or contrast agent: Metal in body: Pacemaker / Automatic Implantable Cardioverter Defibrillators / Implantable Cardioverter Defibrillators (coronary defibrillator), Nervus vagus stimulator, Artificial heart valve (depending on type), Metal clips on cerebral arteries or veins, Metal particles in eye, Port-a-cath, Metal stents, Hydrocephalic pump / insulin pump, Metal implants; f/e screws, prostheses, piercings.
* Claustrophobia, or serious mobility problem (Parkinson, tremors)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate change of composition of cartilage trough imaging marker (dGEMRIC) | 6 months
  To evaluate the techniques for studying proteoglycans content: the delayed gadolinium enhanced magnetic resonance imaging of cartilage (dGEMRIC), after 6 months of treatment with DROGLICAN versus untreated control.

SECONDARY OUTCOMES:
Consumption of Rescue Medication | 6 months
  Use of rescue treatments (Paracetamol or oral NSAIDs excluding COX2 inhibitors)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Vergés, Study Director — Bioiberica
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes